CLINICAL TRIAL: NCT01343628
Title: A Gene by Medication Interaction to the Acute Effects of Alcohol
Acronym: ATX
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to lack of funding
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 13464; K01AA015331 (NIH)
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Alcohol-induced Cue-craving; Alcohol Sensitivity
Keywords: Alcohol, atomoxetine, Strattera, alcohol dependence, alcoholism
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo, Atomoxetine (Placebo Comparator)
  Interventions: Drug: Placebo Comparator
- Atomoxetine, Placebo (Active Comparator)
  Interventions: Drug: Active Comparator: Atomoxetine, Placebo

INTERVENTIONS:
Drug: Placebo Comparator — 16 NET SNP rs 11648486 CC and CT individuals will receive placebo and then after one week washout period, receive atomoxetine. Medications will be given as 2 capsules 1x day for 5 days; active atomoxetine groups will receive 40 mg for 3 days, followed by 80 or 120mg (.91-1.4 mg/kg) on days 4 and 5
  Arms: Placebo, Atomoxetine
Drug: Active Comparator: Atomoxetine, Placebo — 16 NET SNP rs 11648486 CC and CT individuals will receive atomoxetine and then after one week washout period, receive placebo.Medications will be given as 2 capsules 1x day for 5 days; active atomoxetine groups will receive 40 mg for 3 days, followed by 80 or 120mg (.91-1.4 mg/kg) on days 4 and 5.
  Arms: Atomoxetine, Placebo

SUMMARY:
Alcohol dependence, or "alcoholism", affects approximately 14 million Americans. Currently, only three pharmacotherapies (disulfiram, naltrexone, and acamprosate) have been approved for the treatment of alcohol dependence and these medications are, at best, moderately successful. Thus, there is a great need for the examination of other biological systems, which contribute/influence the drug reward/addiction pathways within the brain, such that the discovery of new targets and new pharmacotherapies will be possible. Other biological systems in addition to dopamine, such as serotonin, and norepinephrine (NE) are thought to be important in several aspects of addiction, including reward, craving and depression.

This study will examine the effects of a 5 day course of atomoxetine (a selective NE transporter (NET) inhibitor) (80 mg/day; Strattera or placebo) on alcohol-elicited craving and sensitivity to alcohol. The novelty of this study is that of atomoxetine and the fact that it targets NET, neither of which has heretofore been examined in the context of alcohol dependence. It is hopeful that this study, of 64 total individuals, will provide the PI with sufficient preliminary data to submit a subsequent R01 application to study atomoxetine and the involvement of specific single nucleotide polymorphisms within the NET gene on alcohol-related phenotypes in alcohol dependent and non-dependent populations. The long-term objective of this research is to develop more efficacious treatment interventions for alcohol abuse and dependence.

DETAILED DESCRIPTION:
Design:

NET genotype groups for rs11648486 SNP (CC 61%; CT 33%; TT 4%) (e.g., C/C and C/T) will be compared to one another in a 2 (NET Genotype: C/C vs. C/T & T/T) x 2 (Medication: atomoxetine 80 mg/day (~ vs. placebo) x 3 (Drink: Drink 1, 2, and 3) mixed factorial repeated measures design using PROC MIXED in SAS by calculating difference scores. Of interest are the possible interactions of the NET SNPs and atomoxetine on cue-elicited craving and the rewarding effects of alcohol across trials.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 21 - 45, as verified upon the presentation of a valid, government issued form of ID
* Current DSM-IV diagnosis of alcohol dependence using the Mini International Neuropsychiatric Interview (MINI). Which is a shortened form of the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders or SCID. The MINI will also be used to exclude patients with other diagnoses.
* Participants do not meet DSM-IV criteria for any current (i.e., criteria met at any point in the past 30 days) Axis I disorder (including ADHD treated with medication), other than cocaine dependence or those listed above, that warrants treatment or would preclude safe participation in the protocol
* Not currently take medications that are contraindicated for concurrent use with alcohol;
* No subjects who have trouble reading the English language or visual or hearing problems that may interfere with the collection of data;
* No recurring past history of severe hypertension, glaucoma, hyperthyroidism, circulatory disease, hepatitis, chronic liver disease, ulcer disease, seizure disorder, brain disease, cardiac disease, obstructed bowel, or other current treatment of medical conditions that could determine ineligibility;
* Female subjects must not be breastfeeding and must not be pregnant, as indicated by a pregnancy test that will be conducted immediately prior dispensing of medication.
* Subjects have to have normal EKGs results
* Pulse less than 100 beats per minute
* Participants have to weigh between 125-290; weighing between 125-195 lbs (57 - 88.5 kg)

Exclusion Criteria:

* Significant medical illness (including severe hypertension) as determined by history and/or complete physical examination. (Note: Presence of mild to moderate chronic diseases not otherwise specifically excluded, that are well controlled by medications/interventions will not be considered clinically significant. However the presence of medical disease that is not well controlled will be considered exclusionary.)
* tachycardia
* seizure disorder
* prior history of myocardial infarction
* Clinically significant cardiovascular disease that precludes safe participation
* hepatic or renal impairment; (ie: liver or kidney enzymes > 3x normal limits)
* pregnant
* currently using MAO inhibitors within 14 days

  * narrow angle glaucoma
  * currently taking antidepressants or have taken within the last month
  * currently taking pressor agents such as:
  * Alprenolol
  * Carteolol
  * Levobunolol
  * Mepindolol
  * Metipranolol
  * Nadolol
  * Oxprenolol
  * Penbutolol
  * Pindolol
  * Propranolol
  * Sotalol
  * Timolol
  * Acebutolol
  * Atenolol
  * Betaxolol
  * Bisoprolol[16]
  * Esmolol
  * Metoprolol
  * Nebivolol
  * Carvedilol
  * Celiprolol
  * Labetalol
  * Butaxamine

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2008-01; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Alcohol urge questionnaire | On day 5 of medication
  This questionnaire is used to assess craving. The AUQ consists of eight items related to urge drink that are rated on a 7-point Likert scale with the extremes anchored by "Strongly Disagree" and "Strongly Agree." The AUQ has demonstrated internal consistency and reliability (Bohn et al., 1995).

SECONDARY OUTCOMES:
Biphasic Alcohol Effects Scale (BAES) | On day 5 of medication

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Haughey, PhD, Principal Investigator — University of Virginia
Locations (1):
- Center for Addiction Research and Education, Charlottesville/ Richmond, Virginia, United States